CLINICAL TRIAL: NCT02470611
Title: Effects of 1% Sodium Alendronate in Non Surgical Periodontal Therapy on Clinical and Tomographical Parameters: a Randomized Placebo Controlled 6-month Clinical Trial
Brief Title: Sodium Alendronate in Non Surgical Periodontal Therapy
Acronym: SANSPET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Pontifícia Universidade Católica de Minas Gerais (Other)
Responsible Party: Principal Investigator, Bernardo de Carvalho Dutra, Clinical evaluation and treatment for the effect of image periodontal mechanical non surgical associated with application of topical alendronate sodium a 1% repair periodontal: randomized controlled clinical trial, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE- 22493714.5.0000.5149; 22493714.5.0000.5149 (Other: Ethics committee)
Record Dates: First submitted 2015-06-02; First posted 2015-06-12 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Periodontitis; Bone Resorption
MeSH Terms: conditions — Periodontitis; Bone Resorption | interventions — Alendronate; Diphosphonates

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium Alendronate (Experimental): Adjunctive use of 1% sodium alendronate gel as part of periodontitis treatment
  Interventions: Drug: Sodium alendronate
- Placebo (Placebo Comparator): Adjunctive use of placebo gel as part of periodontitis treatment
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sodium alendronate — After manual quadrant-wise scaling and root planing, at the final treatment appointment the randomized selected periodontal site (showing pocket depth ≥ 5mm, clinical attachment loss > 3mm and proximal bone defects) received 1% sodium alendronate gel
  Other Names: biphosphonates
  Arms: Sodium Alendronate
Other: Placebo — After manual quadrant-wise scaling and root planing, at the final treatment appointment the randomized selected periodontal site (showing pocket depth ≥ 5mm, clinical attachment loss > 3mm and proximal bone defects) received 1% placebo gel
  Arms: Placebo

SUMMARY:
In the past few years, studies have evaluated the effect of systemic use of sodium alendronate, especially in the treatment of structural bone defects caused by periodontal diseases. This study evaluated the effects of non-surgical periodontal treatment associated with the topical application of 1% sodium alendronate on clinical and topographical parameters. Chronic periodontitis patients were recruited for the present study and were monitored at 3 and 6 months after baseline examinations. A placebo gel was used as control.

ELIGIBILITY:
Inclusion Criteria:

* chronic periodontitis
* two contralateral teeth showing periodontal pocket depth ≥ 5mm, clinical attachment loss > 3mm, proximal vertical bone defects, no prosthetic device, without caries lesions, proximal dental contact and lack of premature occlusal contact
* systemically healthy volunteers

Exclusion Criteria:

* need for antibiotic or systemic/local antibiotic use in the previous 3 months
* periodontal treatment in the previous 6 months
* pregnancy or lactation
* immunological disorders or imune suppressive treatments
* diabetes
* smoking
* orthodontic appliances or removable prosthesis
* osteoporosis
* known or suspected allergy to biphosphonates
* systemic use of biphosphonates

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Changes in pocket depth | baseline and 3- and to 6-month evaluations
  Reductions in pocket depth overtime
Changes in clinical attachment level | baseline and 3- and to 6-month evaluations
  Gain in clinical attachment level overtime

SECONDARY OUTCOMES:
Changes in bone defects | Baseline and 6 months
  Reduction in bone defects by bone filling

CONTACTS AND LOCATIONS:
Overall Officials: Fernando O Costa, PhD, Study Chair — Head of Periodontology
Locations (1):
- Dental clinic of pontifical catholic university, Belo Horizonte, Minas Gerais, Brazil